CLINICAL TRIAL: NCT01608360
Title: Intravenous Lidocaine for Effective Pain Relief After Thyroidectomy: a Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Effect of Intravenous Lidocaine on Pain After Thyroidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Kang, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChungAngUH3
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Postoperative Pain
Keywords: Pain; Lidocaine; Intravenous; Thyroidectomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous lidocaine injection group (Active Comparator): Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Interventions: Drug: Intravenous lidocaine injection
- Placebo control group (Placebo Comparator): Patients in Group C (placebo control group) received normal saline intravenous injection
  Interventions: Drug: Intravenous normal saline injection

INTERVENTIONS:
Drug: Intravenous lidocaine injection — Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Other Names: IV lidocaine
  Arms: Intravenous lidocaine injection group
Drug: Intravenous normal saline injection — The patients in Group C (placebo control group) received normal saline intravenous injection
  Other Names: IV saline
  Arms: Placebo control group

SUMMARY:
This prospective randomized study aims to evaluate the effectiveness of intravenous lidocaine injection on the relief of pain in patients undergoing thyroidectomy.

A total 56 patients will be randomized into one of two groups(group C or group I) based on Excel number generation.

Patients in group C will receive normal saline intravenous injection, and patients in group I will receive an intravenous bolus injection of 1.5mg/kg lidocaine followed by a continuous lidocaine infusion of 2mg/kg/hr.

Visual analogue scale pain scores, fentanyl consumption, the frequency at which patients pushed the button(FPB) of a patient-controlled analgesia system, and presence or absence of nausea and vomiting will be recorded at 2,4,8,12,24,48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy

Exclusion Criteria:

* mental change
* allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured using Visual analogue scale at postoperative 2hour | post op 2hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 2hour.

SECONDARY OUTCOMES:
visual analogue scale 4hour | post op 4 hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 4hour.
visual analogue scale 8 hour | Post op 8 hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 8hour.
Visual analogue scale 12hour | Post op 12 hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 12hour.
visual analogue scale 24hour | Post op 24 hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 24hour.
visual analogue scale 48 hour | Post op 48hour
  Patients will be assessed for pain using a visual analogue pain scale(VAS). It is usually a horizontal line, 100mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks ont the line the that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 48hour.
Opioid consumption 2hour | post op 2hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 2hour will be measured.
Opioid consumption 4 hour | Post op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 4hour will be measured
Opioid consumption 8hour | Post op 8 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 8hour will be measured
Opioid consumption 12 hour | Post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 12hour will be measured
Opioid consumption 24 hour | Post op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 24hour will be measured
Opioid consumption 48 hour | Post op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occured. In the case of persistent pain greater than a visual analogue scale(VAS) pain score of 30mm, and additional 50㎍ of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30mm. And sum of delivery from PCA system and and additional opioid fom immediately after operation to post op 48hour will be measured
FPB 2hour | Post op 2 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 2 hour will be measured.
FPB 4hour | Post op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 4 hour will be measured.
FPB 8 hour | Post op 8 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 8 hour will be measured.
FPB 12 hour | Post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 12 hour will be measured.
FPB 24hour | Post op 24hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 24 hour will be measured.
FPB 48 hour | Post op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 48 hour will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kang, Ph.D, Study Chair — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Eun Jin Ahn, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- ChungAng University, Seoul, South Korea

REFERENCES:
- [Derived] Choi GJ, Kang H, Ahn EJ, Oh JI, Baek CW, Jung YH, Kim JY. Clinical Efficacy of Intravenous Lidocaine for Thyroidectomy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. World J Surg. 2016 Dec;40(12):2941-2947. doi: 10.1007/s00268-016-3619-6. PMID 27379388